CLINICAL TRIAL: NCT03714204
Title: Effects of Transcendental Meditation on Physician Burnout and Depression: A Randomized Controlled Trial
Brief Title: Effects of Transcendental Meditation on Physician Burnout and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Loiselle (Other)
Collaborators: Loyola University Chicago (Other)
Responsible Party: Sponsor-Investigator, Marie Loiselle, Researcher, Maharishi International University
Organization: Maharishi International University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1080108
Record Dates: First submitted 2018-10-12; First posted 2018-10-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Burnout, Professional; Depression; Insomnia; Perceived Stress; Resilience
Keywords: academic physician burnout; physician burnout; Intervention to reduce physician burnout; physician depression; physician insomnia; physician stress; Transcendental Meditation; TM
MeSH Terms: conditions — Burnout, Professional; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: The names of individual participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation Group (Experimental): Participants assigned to this group each received the intervention of 5 initial class instructions in the Transcendental Meditation technique, followed by 6 additional classes over the 4-month study period. Group participants were expected to practice the technique for 20 minutes twice per day for 4-months.
  Interventions: Behavioral: Transcendental Meditation technique
- Control Group (No Intervention): Participants assigned to this group served as wait-list controls

INTERVENTIONS:
Behavioral: Transcendental Meditation technique — The TM technique is a simple mental procedure that is categorized in the automatic self-transcending category of meditation practices. It is automatic in that it does not involve any concentration or control. It allows the mental activity to settle down in a spontaneous and natural manner during a process called transcending, or going beyond, until it reaches a state beyond conscious thinking. Correspondingly, the body settles down to a deep state of rest which allows stress to dissolve and the nervous system to rejuvenate The effortless nature of the TM practice coupled with the vast research supporting its efficacy, its systematic standardized teaching program and the fact that it does not involve any belief or change in one's lifestyle made it the choice intervention for this research.
  Arms: Transcendental Meditation Group

SUMMARY:
This research study will examine the effects of the Transcendental Meditation (TM) technique on academic physician burnout, depression, insomnia, perceived stress, and resilience through a mixed methods approach.

DETAILED DESCRIPTION:
Burnout is pervasive among physicians in academia, with costly ramifications for individuals and institutions ($100,000-900,000/faculty replacement). The purpose of this study is to assess, both quantitatively and qualitatively, the effects of the TM technique as an intervention in lowering burnout, depression, perceived stress, insomnia, and to increase resilience in academic physicians.

Research Study Hypotheses Quantitative hypothesis #1: Regular practice of the TM technique by academic physicians for 4 months will reduce symptoms of burnout compared to academic physicians not practicing the TM technique Quantitative hypothesis #2: Regular practice of the TM technique by academic physicians for 4 months will reduce symptoms of perceived stress, insomnia, depression and increase resilience compared to academic physicians not practicing the TM technique.

Qualitative research questions:

1. What are the daily challenges faced by academic physicians and how do they view their ability to handle them?
2. Does regular practice of the TM technique improve their perception of their quality of life with regards to the challenges they face?

Sample Size Estimate There is an effect size of .6225 when using changed scores for treatment and control groups, and their respective standard deviations, from a recent study using the TM technique as the intervention and measuring burnout using the Maslach Burnout Inventory (Elder, 2014). Applying Cohen's power tables for p<.05 to this effect size the number of subjects per group needed is 12. Recruiting 20 subjects per group will allow for 20% attrition.

Study Design Overview The research design is a mixed methods randomized controlled trial (RCT) involving both a treatment and wait-list control group. Quantitative testing will be done three times: pretest followed by posttests at one and four months. The one month posttest is to assess any short term changes as well as a precaution against possible dropouts of either group before the four-month posttest. All subjects will be required to sign an informed consent form prior to participation.

Qualitative data will be gathered through two individual 30-minute semi-structured interviews: the first (entry) before randomization, at the time of the quantitative pretest; and the second (exit) at the 4-month posttest.

The independent variable is instruction in the TM technique, which includes introductory and follow-up sessions to be taught to the treatment group following their pretest and entry interview.

Quantitative data will be analyzed using repeated measures analysis of variance. Qualitative data will be analyzed using a phenomenological approach of identifying main themes and sub themes from the pre and post intervention interviews. The interviews will be the only source of qualitative data. Separate analysis and discussions of quantitative and qualitative data will be merged together to examine their convergence and divergence.

The Institutional Review Board at Maharishi University of Management approved the study in March 2015 followed by the Institutional Review Board at Loyola University Chicago approval in July 2015.

The goal of this study is to see if the intervention alters quantitative measurements of burnout and to understand what kinds of challenges academic physicians face in their daily lives, how they view their ability to handle them, and whether either is transformed during the study period. Although much research has shown symptoms of burnout are largely present among physicians, and a few studies showed promising antidotes, none to date have made use of both quantitative and qualitative data in exploring an intervention for lowering burnout in academic physicians.

This study will employ the advanced convergent mixed methods design which entails collecting both quantitative and qualitative data at pre-and posttest intervals, while adding the advanced feature of an intervention following pretesting.

Study Protocol

* The researcher will oversee all test administration and tracking of subject compliance.
* All study related paperwork and online tests will be managed under appropriate institutional protocol for anonymity and confidentiality. Data will be securely stored appropriately on-line and the hard copies of the consent form kept under lock in the Vice-Dean of Education's office. To further protect the identity of reporting physicians, the identity of the medical school is, and will be, masked in this dissertation and further papers based on this dissertation.

Adverse event reporting: If an adverse event is reported through testing or interviews (and it is a recent issue) it will be reported to the Principal Investigator who will speak to this potential study participant and recommend that they be seen in Employee Health. If the adverse event was suicidal ideation they would be excluded from the study until such time the event was resolved.

ELIGIBILITY:
Inclusion Criteria:

* Have an MD degree
* Be an academic attending physician at the Loyola Chicago School of Medicine or Edward Hines, Jr. VA Hospital
* Commit to attend all required sessions for learning the Transcendental Meditation (TM)technique and monthly follow-ups
* Agree to practice TM twice daily for 20 minutes for the 4-month study period
* Agree to complete both pre-and post-testing (at 1-month and 4-months) including both the entry and exit interviews.

Exclusion Criteria: current suicidal ideation, previous instruction in the TM technique

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory | change from baseline burnout level at four months
  measures burnout level

SECONDARY OUTCOMES:
Beck Depression Inventory | change from baseline depression level at four months
  measures depression level
Insomnia Severity Index | change from baseline insomnia level at four months
  measures insomnia level
Perceived Stress Scale | change from baseline perceived stress level at four months
  measures level of perceived stress
Brief Resilience Inventory | change from baseline resilience level at four months
  measures resilience level

OTHER OUTCOMES:
Personal Interview with researcher | baseline, 4-months
  qualitative assessment

CONTACTS AND LOCATIONS:
Overall Officials: Marie Loiselle, PhD, Study Chair — Outside Researcher; Gregory Gruener, MD, Study Director — Vice-Dean of Education; Carla L Brown, PhD, Principal Investigator — Adjunct Professor
Locations (1):
- Loyola University Stritch School of Medicine, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
all that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be available six months after publication
Access Criteria: To be determined